CLINICAL TRIAL: NCT05111093
Title: Epidural Electrical Stimulation to Restore Hemodynamic Stability and Trunk Control in People With Spinal Cord Injury
Acronym: HemON
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ecole Polytechnique Fédérale de Lausanne (Other)
Responsible Party: Principal Investigator, Jocelyne Bloch, Prof., Centre Hospitalier Universitaire Vaudois
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HemON
Record Dates: First submitted 2021-11-01; First posted 2021-11-08 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- all participants (Experimental): All participants will be provided with the ARC-IM Investigational System (implantable and non-implantable parts)
  Interventions: Device: ARC-IM Investigational System implantation

INTERVENTIONS:
Device: ARC-IM Investigational System implantation — Implantation of a stimulation lead on the low thoracic level of the spinal cord and implantation of a neurostimulator in the abdominal region.

SUMMARY:
The HemON study aims to evaluate the safety and preliminary efficacy of ARC-IM Therapy (Epidural Electrical Stimulation) to improve hemodynamic management and trunk control in people with sub-acute or chronic spinal cord injury (>= 1 month post injury) between C3 and T6 inclusive, who suffer from orthostatic hypotension.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Must provide and sign the Informed Consent prior to any study related procedures
* Spinal cord injury lesion level between C3 and T6 (inclusive)
* SCI ≥ 1month
* Confirmed orthostatic hypotension
* Stable medical, physical and psychological condition as considered by the investigators
* Able to understand and interact with the study team in French or English
* Agrees to comply in good faith with all conditions of the study and to attend all scheduled appointments

Exclusion Criteria:

* SCI related to a neurodegenerative disease
* Diseases and conditions that would increase the morbidity and mortality of spinal cord injury surgery
* The inability to withhold antiplatelet/anticoagulation agents perioperatively
* History of myocardial infarction or cerebrovascular event within the past 6 months
* Other conditions that would make the subject unable to participate in testing in the judgement of the investigators
* Clinically significant mental illness in the judgement of the investigators
* Botulinum toxin vesical and non-vesical injections in the previous 3 months before the enrolment
* Presence of significant pressure ulcers
* Recurrent urinary tract infection refractory to antibiotics
* Presence of indwelling baclofen or insulin pump
* Women who are pregnant (pregnancy test obligatory for woman of childbearing potential) or breast feeding,
* Lack of safe contraception for women of childbearing capacity,
* Intention to become pregnant during the course of the study,
* Other clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, etc.),
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders or dementia of the participant,
* Participation in another study with investigational drug within the 30 days preceding and during the present study,
* Enrolment of the investigator, his/her family members, employees, and other dependent persons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-11-29 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Serious Adverse Events and Adverse Events that are deemed related or possibly related to the study procedure or to the ARC-IM Investigational System | Throughout study, an average of 26 months
  Evaluate the safety of ARC-IM Therapy at supporting management of hemodynamic instability in participants with sub-acute or chronic spinal cord injury suffering from orthostatic hypotension

SECONDARY OUTCOMES:
Orthostatic head-up tilt test (hemodynamic stability assessment) | Baseline ; at 1 - 6.5 - 13 - 26 months after the implantation
  Participant begin by resting in the supine position during which baseline measures are performed. Thereafter, participant is passively moved to upright position using a tilt-table and kept in this position for a maximum of 10 minutes. This test will be performed with and without ARC-IM Therapy. Beat by beat blood pressure is monitored and catecholamine concentrations in the plasma are measured during the tilt-test.
Modified Ashworth Scale (MAS) (spasticity assessment) | Baseline ; at 1 - 13 months after the implantation
  Participants' upper and lower limb spasticity levels (6 points nominal scale) are assessed by rating the resistance of a muscle to a passive range of motion about a single joint. This test will be performed with and without ARC-IM Therapy.
  Scores range from 0 to 5 (0, 1, 1+, 2, 3, 4, 5) with higher scores indicating higher spasticity.
SCIM III (daily life performance assessment) | Baseline ; at 1 - 6.5 - 13 months after the implantation
  The Spinal Cord Independence Measure (SCIM) is a disability score to assess functional activity in participants. Function is assessed in 3 areas of function: self-care (0-20), respiration and sphincter management (0-40) and mobility (0-40). Total score ranges between 0-100, with higher scores reflecting greater functional ability

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyne Bloch, MD, Principal Investigator — CHUV
Locations (1):
- CHUV, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Background] Phillips AA, Squair JW, Sayenko DG, Edgerton VR, Gerasimenko Y, Krassioukov AV. An Autonomic Neuroprosthesis: Noninvasive Electrical Spinal Cord Stimulation Restores Autonomic Cardiovascular Function in Individuals with Spinal Cord Injury. J Neurotrauma. 2018 Feb 1;35(3):446-451. doi: 10.1089/neu.2017.5082. Epub 2017 Nov 21. PMID 28967294
- [Background] Phillips AA, Krassioukov AV. Contemporary Cardiovascular Concerns after Spinal Cord Injury: Mechanisms, Maladaptations, and Management. J Neurotrauma. 2015 Dec 15;32(24):1927-42. doi: 10.1089/neu.2015.3903. Epub 2015 Sep 1. PMID 25962761
- [Background] Squair JW, Phillips AA, Harmon M, Krassioukov AV. Emergency management of autonomic dysreflexia with neurologic complications. CMAJ. 2016 Oct 18;188(15):1100-1103. doi: 10.1503/cmaj.151311. Epub 2016 May 24. No abstract available. PMID 27221275
- [Background] Phillips AA, Warburton DE, Ainslie PN, Krassioukov AV. Regional neurovascular coupling and cognitive performance in those with low blood pressure secondary to high-level spinal cord injury: improved by alpha-1 agonist midodrine hydrochloride. J Cereb Blood Flow Metab. 2014 May;34(5):794-801. doi: 10.1038/jcbfm.2014.3. Epub 2014 Jan 29. PMID 24473484
- [Background] Phillips AA, Elliott SL, Zheng MM, Krassioukov AV. Selective alpha adrenergic antagonist reduces severity of transient hypertension during sexual stimulation after spinal cord injury. J Neurotrauma. 2015 Mar 15;32(6):392-6. doi: 10.1089/neu.2014.3590. Epub 2014 Dec 5. PMID 25093677
- [Background] Phillips AA, Krassioukov AV, Ainslie PN, Warburton DE. Perturbed and spontaneous regional cerebral blood flow responses to changes in blood pressure after high-level spinal cord injury: the effect of midodrine. J Appl Physiol (1985). 2014 Mar 15;116(6):645-53. doi: 10.1152/japplphysiol.01090.2013. Epub 2014 Jan 16. PMID 24436297
- [Background] Krassioukov A, Warburton DE, Teasell R, Eng JJ; Spinal Cord Injury Rehabilitation Evidence Research Team. A systematic review of the management of autonomic dysreflexia after spinal cord injury. Arch Phys Med Rehabil. 2009 Apr;90(4):682-95. doi: 10.1016/j.apmr.2008.10.017. PMID 19345787
- [Background] Phillips AA, Krassioukov AV, Ainslie PN, Warburton DE. Baroreflex function after spinal cord injury. J Neurotrauma. 2012 Oct 10;29(15):2431-45. doi: 10.1089/neu.2012.2507. Epub 2012 Sep 20. PMID 22897489
- [Background] Courtine G, Gerasimenko Y, van den Brand R, Yew A, Musienko P, Zhong H, Song B, Ao Y, Ichiyama RM, Lavrov I, Roy RR, Sofroniew MV, Edgerton VR. Transformation of nonfunctional spinal circuits into functional states after the loss of brain input. Nat Neurosci. 2009 Oct;12(10):1333-42. doi: 10.1038/nn.2401. Epub 2009 Sep 20. PMID 19767747
- [Background] Wagner FB, Mignardot JB, Le Goff-Mignardot CG, Demesmaeker R, Komi S, Capogrosso M, Rowald A, Seanez I, Caban M, Pirondini E, Vat M, McCracken LA, Heimgartner R, Fodor I, Watrin A, Seguin P, Paoles E, Van Den Keybus K, Eberle G, Schurch B, Pralong E, Becce F, Prior J, Buse N, Buschman R, Neufeld E, Kuster N, Carda S, von Zitzewitz J, Delattre V, Denison T, Lambert H, Minassian K, Bloch J, Courtine G. Targeted neurotechnology restores walking in humans with spinal cord injury. Nature. 2018 Nov;563(7729):65-71. doi: 10.1038/s41586-018-0649-2. Epub 2018 Oct 31. PMID 30382197
- [Background] Harkema SJ, Wang S, Angeli CA, Chen Y, Boakye M, Ugiliweneza B, Hirsch GA. Normalization of Blood Pressure With Spinal Cord Epidural Stimulation After Severe Spinal Cord Injury. Front Hum Neurosci. 2018 Mar 8;12:83. doi: 10.3389/fnhum.2018.00083. eCollection 2018. PMID 29568266
- [Background] Aslan SC, Legg Ditterline BE, Park MC, Angeli CA, Rejc E, Chen Y, Ovechkin AV, Krassioukov A, Harkema SJ. Epidural Spinal Cord Stimulation of Lumbosacral Networks Modulates Arterial Blood Pressure in Individuals With Spinal Cord Injury-Induced Cardiovascular Deficits. Front Physiol. 2018 May 18;9:565. doi: 10.3389/fphys.2018.00565. eCollection 2018. PMID 29867586
- [Background] Squair JW, Gautier M, Mahe L, Soriano JE, Rowald A, Bichat A, Cho N, Anderson MA, James ND, Gandar J, Incognito AV, Schiavone G, Sarafis ZK, Laskaratos A, Bartholdi K, Demesmaeker R, Komi S, Moerman C, Vaseghi B, Scott B, Rosentreter R, Kathe C, Ravier J, McCracken L, Kang X, Vachicouras N, Fallegger F, Jelescu I, Cheng Y, Li Q, Buschman R, Buse N, Denison T, Dukelow S, Charbonneau R, Rigby I, Boyd SK, Millar PJ, Moraud EM, Capogrosso M, Wagner FB, Barraud Q, Bezard E, Lacour SP, Bloch J, Courtine G, Phillips AA. Neuroprosthetic baroreflex controls haemodynamics after spinal cord injury. Nature. 2021 Feb;590(7845):308-314. doi: 10.1038/s41586-020-03180-w. Epub 2021 Jan 27. PMID 33505019
- [Background] Darrow D, Balser D, Netoff TI, Krassioukov A, Phillips A, Parr A, Samadani U. Epidural Spinal Cord Stimulation Facilitates Immediate Restoration of Dormant Motor and Autonomic Supraspinal Pathways after Chronic Neurologically Complete Spinal Cord Injury. J Neurotrauma. 2019 Aug 1;36(15):2325-2336. doi: 10.1089/neu.2018.6006. Epub 2019 Mar 6. PMID 30667299
- [Background] West CR, Phillips AA, Squair JW, Williams AM, Walter M, Lam T, Krassioukov AV. Association of Epidural Stimulation With Cardiovascular Function in an Individual With Spinal Cord Injury. JAMA Neurol. 2018 May 1;75(5):630-632. doi: 10.1001/jamaneurol.2017.5055. PMID 29459943
- [Background] Legg Ditterline BE, Aslan SC, Wang S, Ugiliweneza B, Hirsch GA, Wecht JM, Harkema S. Restoration of autonomic cardiovascular regulation in spinal cord injury with epidural stimulation: a case series. Clin Auton Res. 2021 Apr;31(2):317-320. doi: 10.1007/s10286-020-00693-2. Epub 2020 May 13. No abstract available. PMID 32405661
- [Background] Harkema SJ, Legg Ditterline B, Wang S, Aslan S, Angeli CA, Ovechkin A, Hirsch GA. Epidural Spinal Cord Stimulation Training and Sustained Recovery of Cardiovascular Function in Individuals With Chronic Cervical Spinal Cord Injury. JAMA Neurol. 2018 Dec 1;75(12):1569-1571. doi: 10.1001/jamaneurol.2018.2617. PMID 30242310